CLINICAL TRIAL: NCT01737086
Title: Comparing the Efficacy of Two Oral Rehydration Solutions, With or Without the Probiotic Lactobacillus Reuteri DSM 17938 and Zinc, on the Duration and Severity of Acute Gastroenteritis in 6 - 36 Months Old Children in Out-patient Care
Acronym: Profat
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Terminated due to lack of eligible patients.
Sponsor: Umeå University (Other)
Collaborators: BioGaia AB (Industry)
Responsible Party: Principal Investigator, Torbjörn Lind, Associate professor, Umeå University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Profat
Record Dates: First submitted 2012-11-26; First posted 2012-11-29 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Acute Gastroenteritis
MeSH Terms: interventions — Zinc Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ORS with probiotic and zinc (Experimental): Oral rehydration solution with freeze-dried Lactobacillus reuteri DSM 17938 and zinc sulphate
  Interventions: Dietary Supplement: Lactobacillus reuteri DSM 17938 and zinc sulphate
- Standard ORS (Placebo Comparator): Standard oral rehydration solution
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus reuteri DSM 17938 and zinc sulphate
  Arms: ORS with probiotic and zinc
Dietary Supplement: placebo
  Arms: Standard ORS

SUMMARY:
Oral rehydration solution (ORS) is recommended for treatment and prevention of dehydration due to acute gastroenteritis in infants and children. Acute diarrhoea leads to zinc depletion in infants, and zinc is recommended by the World Health Organization in the treatment of acute gastroenteritis in infants and children. However, the efficacy of zinc supplementation to children with acute gastroenteritis in more affluent settings is unclear. Selected strains of probiotics, including L. reuteri ATCC 55730, have been shown in several studies to shorten the duration of diarrhoea by about 24 hours, and also to attenuate symptom severity. If probiotics are given within 60 hours from onset of symptoms the duration can be reduced even more. Lactobacillus reuteri (L. reuteri) has been shown to reduce the duration and severity of acute gastroenteritis in children aged 6-36 months. In these studies L. reuteri was proven to have clinical effect on diarrhoea of both bacterial and viral (rotavirus) origin. In humans, L. reuteri strain DSM 17938 has recently been shown to reduce the duration of watery diarrhoea by 1.2 days among 6-36 mo old Italian children with acute gastroenteritis treated in hospital.

The present, community-based study aims to assess if an ORS with Lactobacillus reuteri DSM 17938 and zinc can be superior or equivalent to ORS without probiotic and zinc in reducing the duration of acute gastroenteritis in children aged 6-36 months, with no, mild or moderate dehydration when introduced early (within 48 hours) after the start of gastroenteritis associated diarrhoea in an out-patient setting.

A prospective, randomized, double blind, controlled study with parallel groups will be performed. Assuming a difference of 25% between groups in the primary outcome of prevalence of diarrhoea 48 hours after start of treatment (80% power, alfa = 5%), and estimating an attrition rate of approximately 15%, the final sample size will be 142 subjects, or 71 subjects in each arm.

Parents contacting the health care telephone enquiry agency, the primary care emergency unit, the paediatric emergency unit, all at the Umeå University Hospital or the well-baby care centres (BVC) in Umeå for advice on their children's gastroenteritis will be informed that they may participate in the present study and they will be given contact information to the research nurse for this activity. A home visit by study personnel will then be done for evaluation of eligibility, information, collection of informed consent and delivery of study product.

Data collection points will be at the recruitment visit in the patient's home, and by telephone on day 7. If the child still has gastrointestinal symptoms on day 5 it will be referred to the primary health care facility or the outpatient clinic of the Department of Paediatrics, Umeå University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* 6 - 36 months of age
* 3 or more loose or watery stools during the past 24 hours
* Available throughout the study period
* Parents or legal guardians are able to give written informed consent to participation in the study.

Exclusion Criteria:

* Diarrhoea with a duration of >48 hours at the time of recruitment.
* Clinical signs of severe dehydration at the time of recruitment or in need of hospitalisation.
* Clinical signs of a coexisting severe acute systemic illness (meningitis, sepsis, pneumonia).
* Primary or secondary immunodeficiency.
* Severe chronic diseases including cystic fibrosis, diabetes mellitus, neurodevelopmental delay or severe gastrointestinal disorders.
* Use of probiotics in the previous 2 weeks before recruitment.
* Use of antibiotics in the previous 2 weeks before recruitment.

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2012-12; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Proportion of children with loose or watery diarrhoea at 48 hours after start of treatment | 48 h after start of treatment

SECONDARY OUTCOMES:
Duration of diarrhoea | 120 hours after start of treatment

OTHER OUTCOMES:
Proportion of children with loose or watery diarrhoea per 24 hour period up to 120 hours after start of ORS treatment. | 120 hours after start of treatment
Number of loose or watery stools per 24 hour period up to 120 hours after start of ORS treatment. | 120 hours after start of treatment
Number of vomiting episodes per 24 hour period up to 120 hours af¬ter start of ORS treatment. | 120 hours after start of treatment
ORS intake during first 24h | 24 hours after start of treatment
Workdays' absence for parents | 7 days after start of treatment
Daycare absence for the child | 7 days after start of treatment
Need of hospitalisation | 7 days after start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Torbjörn Lind, M.D., Ph.D., Principal Investigator — Umeå University
Locations (1):
- Pediatrics, Department of Clinical Sciences, Umeå University, Umeå, Västerbotten County, Sweden